# Evaluating a Digital Peer Mentoring Platform With College Student Populations

NCT05764785

August 2, 2023

# **Study Title**

Evaluating the acceptability, feasibility, and efficacy of a digital peer mentoring platform with college student populations

# **Objectives**

- **Purpose:** The purpose of the study is to assess the acceptability, feasibility, and efficacy of the MentorPRO application with three University of Massachusetts (UMB) student support program-Directions for Student Potential (DSP).
  - o Main outcomes will include attitudes towards the MentorPRO platform, emotional wellbeing (e.g., anxiety, depression), engagement with a third party mental health app, and academic factors (e.g., academic motivation, academic efficacy)
  - o **Research Question 1:** What is the acceptability and feasibility of the MentorPRO mentoring platform?
  - Research Question 2: Does mentoring with MentorPRO demonstrate an impact on academic outcomes (i.e., GPA), engagement with a mental health mobile application, and indices of wellbeing (i.e., mental health, connectedness, academic self-efficacy, and overall wellbeing) among a diverse sample of incoming or first year college students?
- **Study design:** Every student in the DSP program this summer (and meets the study eligibility criteria) will be eligible to participate in the study. Students who opt into participation in research activities will complete 2 brief surveys.
- Study intervention: MentorPRO is a novel application and web platform for mentoring programs that allows students to set goals, track their challenges, and find just-in time resources, while connecting to a mentor for personalized support and progress monitoring. All students in DSP will be matched with a peer mentor. Students will be assigned to getting MentorPRO (intervention condition) or mentoring as usual (control condition), depending on what DSP cohort they are in (a.m. or p.m. classes).
- Study endpoints (clinical trials): All students involved in the DSP summer program will be involved in 6 weeks of academic programming and peer mentoring (June 12th-July 21st), meeting 4 days per week during the summer prior to mentees' first year in college, as well as 3 weeks of post-program peer mentoring (total trial of 9 weeks).

# **Background**

Significance of research question/purpose: Rates of college student distress
have doubled over the past decade, and many of these young people are not
receiving the support they need. There are not enough highly trained supportive
adults in college students' lives (e.g., therapists, counselors, academic advisors,
professors) to prevent mental health, academic, and social challenges or to
directly provide effective interventions. Thus, innovative models of college
student support are necessary to improve this group's overall functioning. Peer

- mentoring is one method of providing direct support to students, task-shifting day-to-day student challenges to peers, allowing academic advisors and other supportive adults the time to focus on more pressing concerns. Over the recent years, technology-enhanced and technology-delivered interventions for academic, mental health, and other outcomes have also been gaining popularity and have recently entered the mentoring space. Research is needed to understand the efficacy of technology-enhanced mentoring models to support university students, particularly those of vulnerable populations.
- Preliminary data: The MentorPRO application was examined in previous program evaluations with a first year college student mentoring initiative at a university in the northeastern United States. Results of these studies demonstrated that MentorPRO was both acceptable and feasible (Werntz et al., 2023). Propensity score matching with students at the same mentoring initiative indicated that greater engagement with peer mentors and greater engagement with a student support smartphone app, MentorPRO, are significantly related to better student academic outcomes and perceived wellbeing (Werntz et al., in preparation).
- Background literature with references: A growing number of researchers have suggested more effectively leveraging more experienced peers to support first year students (Wilson & Gore, 2013). Assigning peer mentors through formal programs can help to address the fact that more marginalized students often struggle to recruit college-based mentors on their own (Gowdy et al., 2020; Hagler et al., 2021). Unfortunately, most peer mentoring programs emphasize nonspecific, relational approaches, and provide uneven training and oversight (Burton et al., 2022; Christensen et al., 2020), resulting in small to non-existent effects on students' psychological, academic, and behavioral difficulties (Christensen et al., 2020; DuBois et al., 2011; Raposa et al., 2019). A meta-analysis of 48 youth mentoring studies showed that the overall effect size of programs that target specific goals are double that of non-specific relational approaches overall, and three times more effective in improving academic, psychological, and social functioning (Christensen et al., 2020). Moreover, research on cross-age peer-mentoring programs emphasize the importance of peer training; peer mentors have moderate effects on mentees' outcomes overall (g=0.45), but there are no measurable effects (g=0.03) when there is low oversight (Burton et al., 2022). Particularly given the enormous potential of peer mentors to bridge growing gaps in student support, these studies suggest a need for college peer-mentoring approaches that (a) provide sufficient training and support of mentors (b) track and support students' early challenges; (c) are grounded in targeted, goal-focused, evidence-based approaches; and (c) are integrated with campus reporting systems. Moreover, mobile platforms can help to support and scale these approaches. Based on these principles, MentorPRO was developed in partnership with researchers, university staff, and students. Early evaluations of MentorPRO demonstrated that MentorPRO was both acceptable (Wertnz et al., 2023) and feasible (Werntz et al., 2023). Propensity score matching with students at the same mentoring initiative indicated that

greater engagement with peer mentors and greater engagement with a student support smartphone app, MentorPRO, are significantly related to better student academic outcomes and perceived wellbeing (Werntz et al., in progress).

Although preliminary evaluations have shown the promise of the MentorPRO platform for promoting positive student outcomes, additional research is needed with other student populations, especially disadvantaged student populations. The university in which data was collected for Werntz et al. (2023) is a predominately-white institution (43.8% white students, 57.0% white faculty, 59.8% white staff as of Fall 2021) with highly competitive academics (75% of the first year class had a high school GPA above 4.1/5). Therefore, it might be that risk is less pronounced than other universities. Additional research is needed to understand if MentorPRO holds similar efficacy at colleges and universities with more diversity and/or where students are at greater risk of dropping out. Researching the implementation of MentorPRO in the already-established CLA First, DSP, and SSS programs will allow researchers to measure the impact on student outcomes across more disadvantaged groups that are at higher risk.

## **Study Population**

- The current study will include an evaluation of the MentorPRO app with a program at UMB:
  - o The <u>Directions for Student Potential</u> summer program (<u>DSP</u>) invites academically-vulnerable incoming students to participate in a summer preparation course (the summer before their first year). Students are matched with peer mentors who are former DSP students.
- Inclusion and exclusion criteria:
  - o The inclusion criteria for the current evaluation includes:
    - Being 18 years of age or older
    - Being a current member of DSP
    - Can speak, read, and write in English
    - Has access to a smartphone
  - o **Inclusion of vulnerable populations**: All participants will be UMB undergraduate students. Participants will *not* include any prisoners, pregnant women (that we are aware of), anyone under the age of 18, or adults unable to consent.

#### **Study Duration**

 All students involved in the DSP summer program will be involved in 6 weeks of academic programming and peer mentoring (June 12th-July 21st), meeting 4 days per week during the summer prior to mentees' first year in college, as well as 3 weeks of post-program peer mentoring (total trial of 9 weeks).

 Investigators will be collecting data between June 2023 and August 2023. After data has been collected, investigators are expected to run analyses, provide reports to partnering programs, and write up manuscripts through summer of 2024.

# **Number of Participants**

- The DSP Summer program serves up to 300 incoming students.
- At the end of the study, mentors will also be recruited for participation. The estimated number of mentors is 10.
- The number of students who opt into the research activities are expected to be lower than the total number of students in the program.

## **Setting**

- Sites/locations:
  - o The current study will include an evaluation of the MentorPRO app with DSP.
  - o Participants will be involved in an already-established mentoring program through UMB, and will be recruited for additional evaluation efforts from the already-established program.
  - o All data collection will occur via online platforms. MentorPRO collects various data points from users directly through the app, including but not limited to: responses to in-app surveys and check-ins, in-app chat messaging, and app engagement. For the students who opt into additional research activities, all surveys will be conducted via UMass Boston's Qualtrics.
- Prior approvals: N/A
- External IRB/ethics review: N/A
- Local permissions/local context: N/A

## **Recruitment Methods**

- Recruitment process: During the DSP programming, DSP staff will hand out postcards that has information about the study and a QR code to sign up (Qualtrics). The Qualtrics link will have (in order): an informed consent, an eligibility screener, and if eligible, the pre-intervention survey (Time 1; T1).
  - o Students will have time to ask questions, and any questions in which program staff cannot answer will be escalated to the research team. Individuals will also be provided the contact information of the study Principal Investigator (Dr. Jean Rhodes) in the consent form so that they can ask any questions before consenting, if relevant.
- Recruitment materials: During the DSP programming, DSP staff will hand out postcards that have information about the study and a QR code to sign up on (Qualtrics). See attached.

- Screening for eligibility: All interested participants will be required to take a brief eligibility screening via Qualtrics. If a student does not meet the criteria, the Qualtrics survey will close and not let them proceed with the study. The only inclusion criteria for the current evaluation includes:
  - o 18 years of age or older
  - o Being a current member of DSP
  - o Can speak, read, and write in English
  - o Has access to a smartphone

0

## **Procedures Involved**

- Study procedures:
  - o Student mentees:
    - All interested participants will read and sign an informed consent, after having time to ask questions to program staff and the research team. Then, they will complete an eligibility screener, and if eligible will complete the rest of the baseline survey.
    - Interested participants will then be prompted to take the first survey after consenting to the study (T1). Students will complete the DSP course for 6 weeks, and will receive peer mentoring during that time. For 3 weeks after the course, students will be able to contact their peer mentor with questions. At the end of the 9-week trial, students will receive a final survey (T2). The eligibility screener, informed consent, and the surveys will be administered via a Qualtrics link. At the conclusion of their participation, all participants will receive a debriefing statement explaining the study and where to find additional resources if needed.
    - Students will be assigned to the intervention or control condition based on what DSP cohort they are part of (a.m. or p.m. classes the a.m. cohort will be assigned to the intervention/MentorPRO condition, while the p.m. cohort receives mentoring as usual).
    - Mentors will be matched with students who are assigned to both conditions, and therefore all mentors will receive all training materials. In addition to the training in program policies and relationship building provided to program peer mentors, all mentors will undergo training designed by the research team. Mentors will complete a brief orientation to the MentorPROUMB technology, followed by a 30-min interactive online course on providing supportive accountability, through MentorPRO UMB Academy which includes "knowledge checks" to ensure mentors are engaged and understanding the material and tracks progress to ensure course completion. Finally, mentees will be given access to an online orientation to MentorPRO UMB, which walks them

- through instructions about how to download and use the app. All study participants (mentors and student mentees) will have access to tech support within 24 hours from Academic Web Pages for any questions or issues that arise.
- Students in the intervention condition may be recommend a third-party mental health app (Healthy Minds Program; HMP) and be provided supportive accountability (i.e., encouragement, nudges, etc) from their mentor to promote consistent active engagement with HMP. Mentors will have three handouts for HMP; one for how to talk about HMP with students, one for how to provide support to students, and one for students that instructs them on how to download the app. Please see attached handouts (3). Data on students' engagement with HMP will be provided weekly from the Healthy Minds team (exported from Amazon Web Services by the research team) and distributed to the appropriate mentor weekly to inform individual supportive accountability practices.
- All study measures administered via Qualtrics can be found attached. The following data will also be requested from academic records at UMB:
  - Pre-matriculation/High school GPA
  - Course load/credits for fall '23 semester
- Additional data sources:
  - HMI app data
    - o Engagement
    - o Responses to in-app questionnaires
  - MentorPRO app data
    - o Engagement
    - o Responses to in-app questionnaires
  - Mentors' engagement in MentorPRO Academy training courses

#### o Mentors:

 At the end of the 9 weeks, mentors will be recruited to provide feedback. Interested mentors will fill out an eligibility screener, and, if eligible, an informed consent form, brief demographics survey, and short feedback survey (all through Qualtrics). See the attachment for all mentor measures.

#### • Payment/incentives:

- o Students will receive \$50 for the first survey and \$50 for the final survey. Therefore, if they complete all three surveys, they can earn up to \$100. Payment will be administered to participants via Tango Gift Cards at the end of the study.
- Mentors will receive \$10 for the feedback survey. Payment will be administered to participants via Tango Gift Cards at the end of the study.

- o Because students in the **MentorPRO** condition are being asked to do additional tasks (compared to students who are not in the MentorPRO condition), students in the MentorPRO condition will be allowed to participate in a raffle for a MacBook Air (valued at \$899) for the use of MentorPRO. Students in the MentorPRO condition are being asked to use MentorPRO and the Healthy Minds every day, resulting in up to 35 minutes of effort a day. Given this effort, we feel that this opportunity is adequate compensation. If all participants earn a similar number of chances, the probability of winning the MacBook Air is 1/25 (4 % chance).
  - 5 entries for messaging with their Peer Navigator each week through Aug 11
    - Now through July 28
    - July 28-Aug 4
    - Aug 5 Aug 11
  - 1 entry for each Check-In before Aug 11
  - 5 entries downloading/installing/following directions to get onto Healthy Minds
  - 1 entry for every day of Healthy Minds use after initial use Students in the MentorPRO condition who have already consented to the study will be informed of the raffle via text, email, and/or phone call and will be given the raffle information, including the attached PDFs (explaining the raffle, and how to get started with Healthy Minds). Questions will be answered by research staff.

# **Data Analysis**

- **Data analysis:** The data will be analyzed both quantitatively and qualitatively. The procedures are outlined below to address each of the research questions:
  - o Research Question 1: What is the acceptability and feasibility of the MentorPRO mentoring program?
    - Recruitment, retention, and adherence to the MentorPRO mentoring program and application will be evaluated to determine the acceptability and feasibility of the program.
    - Acceptability of MentorPRO will also be assessed through open-ended questions and surveys commonly used to evaluate online programs.
    - Qualitative analyses will be conducted to evaluate the level of participants' engagement with mentors via the in-app chat messaging feature.
    - Mentors' responses to survey questions will examine initial mentor feasibility and acceptability of MentorPRO.
  - Research Question 2: Does mentoring with MentorPRO demonstrate an impact on efficacy for student academic outcomes (i.e., GPA) and indices of wellbeing (i.e., mental health, connectedness, academic self-efficacy,

and overall wellbeing) among a diverse sample of incoming or first year college students?

- Quantitative analyses will be conducted to determine whether level of engagement with mentors and the app (e.g., via frequency of in-app chat messaging, frequency of in-app survey completion and check-ins) relates to changes in academic outcomes and indices of wellbeing, as well as to broadly model how these domains change over the course of students' participation.
- Group comparisons will be conducted to examine if there are differences in final mental health and wellbeing measures across groups (intervention and control). Baseline demographics and wellbeing indices will be used as covariates in analyses.
- o Exploratory analyses will also be conducted on the data to examine whether other trends or patterns emerge from the data.

#### Data integrity:

 In order to ensure quality control of the data collected via the Qualtrics survey, participants will be prevented from submitting multiple responses by enabling this feature within Qualtrics. Data will be checked for missingness.

# Risks to Participants

- The potential risks are minimal for this research project, as a majority of the procedures in this study that participants will be exposed to are no more a risk than what individuals encounter on a daily basis. Participants may experience some emotional discomfort related to assessment questions, which ask about academic performance, emotional wellbeing, and emotional and social functioning. However, asking these questions is pertinent to the goals of this study in order to compare changes on variables throughout the intervention.
- Participants can skip any questions on the survey that they would prefer not to answer or stop participating at any time, which will be made clear on the informed consent and during the survey completion process.
- There is a slight risk for breach of confidentiality as participation in the research is dependent on membership in a UMB program.
- Researchers will have access to identified data from the MentorPRO application and surveys to match data across datasets and for the purpose of compensating individuals for their study participation. All other researchers will receive de-identified matched data. All analyses will be run on de-identified datasets and findings will be reported in aggregate form.
- In the informed consent and debriefing form, there will be information on where to find resources for emotional support at UMB in the rare case that any of the participants need additional support.

# **Potential Benefits to Participants**

 Participants will not directly benefit from this study. However, findings from this study will inform how MentorPRO can be used to support students in the best way possible. Findings will reveal what aspects of MentorPRO work well, and where improvement might be needed for future implementations that the student may be involved in.

### **Resources Available**

- All members of the research team are either professionals or graduate-level students in psychology, all with research experience and some with clinical experience.
- The Principal Investigator (Dr. Jean Rhodes) is an expert in mentoring practices. Rhodes has dedicated her career to investigating the ways in which mentoring can be revolutionized to improve outcomes for all involved. She founded the Center for Evidence-Based Mentoring at UMB and is the co-founder of MentorPRO.
- The PI (Dr. Jean Rhodes) and Co-PI (Dr. Alexandra Wertnz) both have their doctorate in clinical psychology.
- All researchers involved in this project have certificates in the CITI ethics training and will read the IRB protocol to ensure understanding. Regular team meetings will be held to discuss the project and provide any updates needed to retain ethical practices and adherence to the protocol.
- In the informed consent, assent, and debriefing forms, participants will be provided with resources they can access if they need additional emotional support - including the university counseling centers and the IRB board at UMB if they have further questions regarding the research.

#### **Consent Process**

- All students in the program will be invited to participate in the research project
  via the outlined recruitment methods. From there, all interested participants will
  read and sign an informed consent. The consent form will be administered via a
  Qualtrics link, in which participants cannot move forward with the study until
  they have consented.
- To protect participants, all interested students will have time to ask questions to program staff and the research team before consenting. Further, the informed consent will make it clear that participation in the research activities (surveys) are optional, any survey questions can be skipped, and they can stop participation at any time without negative consequences to their academic standing or participation in the associated UMB program.
- The informed consent will also have resources provided in the rare case that additional support is needed throughout or after participation.
- Please see attached for a copy of the informed consent and debriefing forms.
- No incomplete disclosure nor deception will be used in this study.

# **Vulnerable Populations**

- All participants in the study will include UMB students.
- The majority of the research team does not teach, supervise or have the ability to influence participants' grades, academic success, or professional advancement.
- The PI (Dr. Jean Rhodes) teaches at UMB in the psychology department, and it is possible that one of the participants may end up as her student for courses and/or advisee for activities outside of the program. However, while the PI will have access to identifiable data from the Qualtrics survey, other research team members will be tasked with handling this identifiable data for the purpose of merging the survey data across time points into one dataset and for de-identifying the dataset for other research team members to access.
- In the informed consent and debriefing form, it will be made clear to participants that neither their participation in the research project nor their responses to survey items will affect grades, academic success, or professional advancement. Participants will also be informed that they can stop participating at any time or skip any questions on surveys if they wish to not respond.

•

- It will be made clear to participants during recruitment, the informed consent process, and debriefing that choosing to not participate in the additional research activities (or stop after participation has already begun) will not affect their membership nor performance in the associated UMB program.
- If participants choose to stop participation, it will be clear in the informed
  consent that they should stop the survey and close the browser. If they choose to
  not have any of their data used for the study, they will be informed to contact
  Megyn Jasman to have the survey data removed from the study (survey data will
  be deleted).

# **Provisions to Protect the Privacy Interests of Participants**

- As part of their involvement in the already-established program at UMB (DSP),
   MentorPRO will collect data on their engagement with the app, communications
   through the app, and any surveys or related questions answered within the app.
   This data is stored on the MentorPRO admin dashboards, which are only
   accessible to the MentorPRO team (which includes 4 of the researchers Rhodes,
   Werntz, Hersch, and Jasman) and is password protected.
- Raw survey data collected for this research project will have identifiers (name and email), which will allow matching between survey responses and MentorPRO data, as well as academic records. All data will be stored in UMB's OneDrive under password protection. Only specified researchers will have access to identified datasets. All analyses will be run on de-identified datasets and presented in aggregate form.
- Data on students' engagement with a third-party mental health app (HMP) will be provided weekly from the Healthy Minds team (exported from Amazon Web Services by the research team) and distributed to the appropriate mentor weekly

to inform individual supportive accountability practices. More specifically, once the identified engagement data is downloaded by the research team, it will be uploaded to a password protected UMB OneDrive folder that the entire research team has access to. From there, the research team will organize the data and place the identified data in a password-protected folder specific to the mentor (1 for each mentor). Data will be identified so that mentors know which students to provide supportive accountability to. However, mentors will only get engagement data in their folders for the students in which they are working with. Once completed, the researcher will immediately delete the downloaded file from their personal machines. DSP staff will inform mentors when their folders have been updated with such information. DSP program staff may also see identified HMP engagement data, as they will have access to the mentor's folder to ensure mentors receive the materials. However, DSP staff will not have access to any identified survey data.

 Participants will be informed on these steps to maintain their privacy in the informed consent, while leaving time to ask questions.

# **Data Confidentiality**

- Identifiers are already collected for academic records and MentorPRO.
- Identifiers will be collected via Qualtrics to allow matching datasets (between surveys, MentorPRO data, and academic records). The research team will have access to identified data only until data have been matched across sources.
- Identifiers will be stored on a password protected computer by the research team. Identified data will only remain identified until the data from various sources has been merged. Once data has been merged, the full dataset will be de-identified. A list of participant IDs and identifiers will be kept separate from the individual responses after the dataset is de-identified. Data and the list of participant IDs/participant identifiers will be stored in UMB's OneDrive under password protection.
- De-identified data may be stored for use in future studies without notifying participants. Participants will be informed of this in the informed consent and debriefing form.
- Data on students' engagement with a third-party mental health app (HMP) will be provided weekly from the Healthy Minds team (exported from Amazon Web Services by the research team) and distributed to the appropriate mentor weekly to inform individual supportive accountability practices. More specifically, once the identified engagement data is downloaded by the research team, it will be uploaded to a password protected UMB OneDrive folder that the entire research team has access to. From there, the research team will organize the data and place the identified data in a password-protected folder specific to the mentor (1 for each mentor). Data will be identified so that mentors know which students to provide supportive accountability to. However, mentors will only get engagement data in their folders for the students in which they are working with. Once completed, the researcher will immediately delete the downloaded file from

their personal machines. DSP staff will inform mentors when their folders have been updated with such information. DSP program staff may also see identified HMP engagement data, as they will have access to the mentor's folder to ensure mentor's receive the materials. However, DSP staff will not have access to any identified survey data.

MentorPRO will continue to store MentorPRO data even after participants finish
or stop participating in the study, which participants will be made aware of in the
informed consent.

## **Data (and Specimen) Banking for Use in Future Studies**

- De-identified data may be stored for use in future studies without notifying participants. Participants will be informed of this in the informed consent and debriefing form.
- All de-identified data will be stored by the research team on password-protected computers and UMB's OneDrive.

#### **Sharing of Results with Participants**

• There are no plans to explicitly report findings directly to participants.

#### **Economic Burden to Participants**

• There is no expected economic burden to participants.

#### **Withdrawal of Participants**

• n/a

#### **Community-Based Participatory Research**

• n/a

#### **Compensation for Research-Related Injury**

• n/a

#### Provisions to Monitor the Data to Ensure the Safety of Participants

• n/a

#### **Multi-Site Research**

• n/a

#### References

Burton, S., Raposa, E. B., Poon, C. Y. S., Stams, G. J. J. M., & Rhodes, J. (2022). Cross-age peer mentoring for youth: A meta-analysis. *American Journal of Community Psychology,* 70(1-2), 211-227. https://doi.org/https://doi.org/10.1002/ajcp.12579

Christensen, K. M., Hagler, M. A., Stams, G., Raposa, E. B., Burton, S., & Rhodes, J. E. (2020). Non-specific versus targeted approaches to youth mentoring: A follow-up meta-analysis. *Journal of Youth and Adolescence*, *49*, 959–972. https://doi.org/10.1007/s10964-020-01233-x

DuBois, D. L., Prtillo, N., Rhodes, J. E., Silverthorn, N., & Valentine, J. C. (2011). How effective are mentoring programs for youth? A systematic assessment of the evidence. *Psychological Science in the Public Interest*, *12*(2), 57–91. https://doi.org/10.1177/1529100611414806

Gowdy, G., Miller, D. P., & Spencer, R. (2020). Expanding and deepening our understanding of which young people are most likely to have an informal mentor. *Children and Youth Services Review, 108*. https://doi.org/10.1016/j.childyouth.2019.104490

Hagler, M. A., Christensen, K. M., & Rhodes, J. E. (2021). A longitudinal investigation of first-generation college students' mentoring relationships during their transition to higher education. *Journal of College Student Retention: Research, Theory & Practice*. https://doi.org/10.1177/15210251211022741

Raposa, E. B., Rhodes, J., Stams, G.J., Card, N., Burton, S., Schwartz, S., Sykes, L.Y., Kanchewa, S., Kupersmidt, J., and Hussain, S. (2019). The effects of youth mentoring programs: A meta-analysis of outcome studies. *Journal of Youth and Adolescence*. https://doi.org/10.1007/s10964-019-00982-8

Werntz, A., Jasman, M., Simeon, K., Gunasekaran, H., Yowell, C., & Rhodes, J. (2023). Implementation of a technology-enhanced peer mentor referral system for first-year university students., Journal of Technology in Behavioral Science. <a href="https://doi.org/10.1007/s41347-023-00303-8">https://doi.org/10.1007/s41347-023-00303-8</a>

Werntz, A., Deng, Y., Jasman, M., Yowell, C., & Rhodes, J. E. (in progress). Effects of a technology-enhanced university peer mentoring program on first semester academic and wellbeing outcomes: A propensity score matching analysis.

Wilson, S., & Gore, J. (2013). An Attachment Model of University Connectedness. *The Journal of Experimental Education*, 81(2), 178-198. https://doi.org/10.1080/00220973.2012.699902